CLINICAL TRIAL: NCT05356741
Title: A Phase 1, Multicenter, Open-Label, First-in-Human Study of the Safety and Pharmacokinetics of VIR-5818 Alone and in Combination With Pembrolizumab in Participants With Locally Advanced or Metastatic HER2-Expressing Cancers
Brief Title: To Access the Safety and Effects of Intravenous Administration of VIR-5818 Alone and in Combination With Pembrolizumab in Adult Participants With Locally Advanced or Metastatic HER2-Expressing Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIR-5818-V101; MK-3475-D14 (Other: Merck Sharp & Dohme LLC); KEYNOTE-D14 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic HER2-Expressing Cancers
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 (dose escalation) (Experimental): Participants will receive single-agent VIR-5818
  Interventions: Drug: VIR-5818
- Part 2 (dose escalation) (Experimental): Participants will receive VIR-5818 plus pembrolizumab
  Interventions: Drug: VIR-5818; Drug: pembrolizumab
- Part 3 (dose expansion) (Experimental): Participants will receive single-agent VIR-5818
  Interventions: Drug: VIR-5818
- Part 4 (dose expansion (Experimental): Participants will receive VIR-5818 plus pembrolizumab
  Interventions: Drug: VIR-5818; Drug: pembrolizumab

INTERVENTIONS:
Drug: VIR-5818 — Administered as IV infusion
Drug: pembrolizumab — Administered as IV infusion
  Other Names: KEYTRUDA®
  Arms: Part 2 (dose escalation); Part 4 (dose expansion

SUMMARY:
This first-in-human (FIH) Phase 1 open-label multicenter dose-escalation and dose-expansion study is designed to evaluate the safety, pharmacokinetics, and preliminary activity of VIR-5818 (Formerly AMX-818) as a single agent and in combination with pembrolizumab in participants with HER2+ tumors across multiple tumor types. The study will be conducted in four parts:

* Part 1 (dose escalation): Single-agent VIR-5818
* Part 2 (dose escalation): VIR-5818 plus pembrolizumab
* Part 3 (dose expansion): Single-agent VIR-5818
* Part 4 (dose expansion): VIR-5818 plus pembrolizumab

The total length of the study, from screening of the first participant to the end of the study, is expected to be approximately 52 months.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent by the participant (or legally acceptable representative if applicable)
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Diseases under study, prior lines of therapy, and human epidermal growth factor receptor 2 (HER2) status, per local tests

Exclusion criteria:

* Significant cardiopulmonary disease and recent cardiac events
* History of major organ autoimmune diseases
* Acute or chronic infections

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 645 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2027-08-16 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity - Part 1 and Part 2 | Up to approximately 21 days (Part 1) and 42 days (Part 2)
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)- Parts 1, 2, 3, and 4 | Up to approximately 55 months
Objective Response Rate (ORR) - Part 3 and Part 4 | Up to approximately 55 months
  ORR defined as a Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
Duration of Response (DOR) - Part 3 and Part 4 | Up to approximately 55 months
  DOR defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per RECIST v.1.1.

SECONDARY OUTCOMES:
ORR - Part 3 and Part 4 | Up to approximately 55 months
  ORR defined as defined as a Complete Response (CR) or Partial Response (PR) per Immune Response Evaluation Criteria in Solid Tumors (iRECIST).
DOR - Part 3 and Part 4 | Up to approximately 55 months
  DOR defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per iRECIST.
Pharmacokinetics (PK) parameter: Area under the concentration-time curve (AUC) | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
PK parameter: Maximum plasma concentration (Cmax) | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
PK parameter: Minimum serum concentration (Cmin) | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
PK parameter: Clearance (CL) | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
PK parameter: Volume of distribution at steady-state (Vss) | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
PK parameter: Accumulation ratio | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
PK parameter: Half-life (t1/2) | Predose, intermediate timepoints at multiple cycles (1 Cycle = 21 days) up to approximately 55 months
Incidence of anti-drug antibodies (ADAs) to VIR-5818 | Multiple timepoints at specified cycles (1 Cycle = 21 days) up to approximately 55 months
All parts: Disease control rate (DCR) | Up to approximately 55 months
  defined as CR+PR+ Stable Disease (SD) per RECIST v 1.1

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (2):
  - Investigational site number #100, Melbourne, Victoria
  - Investigational site number #101, Randwick
- Investigational site number #150, Toulouse, France
- Investigational site number #200, Porto, Portugal
- Spain (6):
  - Investigational site number #255, Barcelona
  - Investigational site number #251, Barcelona
  - Investigational site number #254, Madrid
  - Investigational site number #252, Madrid
  - Investigational site number #250, Pamplona
  - Investigational site number #253, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: Yes